CLINICAL TRIAL: NCT04877626
Title: Assessment of the Therapeutic Efficacy and Tolerability of the Artesunate/Amodiaquina Combination and Artemether/Lumefantrine Combination, the Standard Treatment Recommended by the Ministry of the Social Protection in Colombia for the Treatment of Uncomplicated P. Falciparum Malaria in the Department of Chocó (Colombia)
Brief Title: Assessment of the Therapeutic Efficacy and Tolerability of the Artesunate/Amodiaquina Combination and Artemether/Lumefantrine Combination, Treatment of Uncomplicated P. Falciparum Malaria in the Department of Chocó (Colombia)
Acronym: UNAL MALARIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad Nacional de Colombia (Other)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Treatment malaria in Colombia
Record Dates: First submitted 2010-06-24; First posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: P. Falciparum Malaria
Keywords: uncomplicated P. falciparum malaria; Colombia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AQ+AS (Active Comparator): Group 1 received the combination AQ+AS (COARSUCAM®) which was administered orally at an initial dose of 2 tablets (200 mg AQ/540 mg AS) followed by 2 additional doses of 2 tablets at 24 and 48 hours (6 tablets in 48 hours).
  Interventions: Drug: Artemeter plus lumefantrina vs artesunato plus amodiquina
- AM+L (Active Comparator): Group 2 received the combination Artemeter+lumefantrina (COARTEM®) administered orally at an initial dose of 4 tablets (80 mg artemeter/480 mg lumefantrina) followed by 5 additional doses of 4 tablets at 8, 24, 36, 48, and 60 hours (24 tablets in 60 hours)
  Interventions: Drug: Artemeter plus lumefantrina vs artesunato plus amodiquina

INTERVENTIONS:
Drug: Artemeter plus lumefantrina vs artesunato plus amodiquina — Group 1 received the combination AQ+AS (COARSUCAM®) which was administered orally at an initial dose of 2 tablets (200 mg AQ/540 mg AS) followed by 2 additional doses of 2 tablets at 24 and 48 hours (6 tablets in 48 hours).
  Group 2 received the combination Artemeter+lumefantrina (COARTEM®) administered orally at an initial dose of 4 tablets (80 mg artemeter/480 mg lumefantrina) followed by 5 additional doses of 4 tablets at 8, 24, 36, 48, and 60 hours (24 tablets in 60 hours)

SUMMARY:
Background: Malaria by P falciparum is a public health problem in more than 100 municipalities of Colombia. The country is using the artemether+lumefantrine (AM+L) fixed combination for uncomplicated P falciparum malaria but it is ideal to have different types of formulations with similar efficacy that may be used in diverse circumstances. One alternative of treatment is using preparations containing artesunate and amodiaquine (AS+AQ) in fixed combination, which can be given in a simpler dosing regimen. In order to assess the efficacy of that combination in an area with suspected risk of resistance to amodiaquine an open controlled clinical trial was carried out in Colombia. Methods: The study was done in Choco, a high endemic area for malaria by P falciparum, from August 2008 and September 2009. Patients diagnosed with uncomplicated malaria (n=210) malaria were randomized in two arms, one receiving AS+AQ and the other AM+L. The main clinical results was parasitological cure, i.e. a negative blood smears, that was assessed, for both groups, at days 1, 2, 3, 7, 14, 21 and 28 after the onset of treatment. Results: There were no losses at follow up. The mean age of the enrolled study subjects was of 37.5 years without differences between study arms. Both therapies were very well tolerated in general. The efficacy for AS+AQ was 100%, and 99% for AM+L (p>0.1). In average, patients in the AS+AQ arm became negative for P falciparum parasites and gametocytes earlier than those at the AM+L arm. Blood smears became negative after one day of treatment with AS+AQ and after two days of treatment with AM+L. Gametocytes disappeared after 2 days of treatment in the AS+AQ arm compared to 4 days in the AM+L arm. Conclusions: In this study, the efficacy of the AS+AQ combination was similar to that of the AM+L. This finding do not support the hypothesis that there is a level of resistance to amodiaquine that prevents its use combined with artemisinin derived.

DETAILED DESCRIPTION:
Design: An open-labeled, randomized and controlled clinical trial with follow-up in days 1, 2, 3, 4, 7, 14, 21 and 28 was carried out in adult patients with uncomplicated P. falciparum malaria. This type of study has been validated by PAHO and has been used by the Amazon Network for the Surveillance of Antimalarial Drug (RAVREDA) to evaluate the efficacy of antimalarial treatment in the Americas region. This study is a simplified version with monthly follow-up by a Data Safety Monitoring Board (DSMB) of the status of therapeutic failures to assure that the study progress does not result unethical.

Study area: The study area was in Department of Chocó, which is located west in the Pacific region of the country, has an approximate extension of 47,000 Km2, equivalent to 4% of the country's total extension. Chocó has 31 Municipalities for a total of 454,030 inhabitants, according to the 2005 Survey. From this population, 90% is black, 6% mulatto or white, and the remaining 4% natives. The great part of the population has its settling in the river and sea zones, which constitutes an important aspect to consider in communications, culture and socioeconomic development of the region. The temperature ranges between 26º and 30ºC. Patients were recruited from two municipalities, Quibdo and Tado.

Inclusion Criteria. Age > 18 years, fever (axillary temperature >37.5º C) or history of fever during the prior 48 hours in absence of another obvious cause (such as pneumonia, otitis media), a non-mixed P. falciparum infection with 250 and 100,000 asexual parasites/µl to be determined by a thick film or thick film and blood smear microscopic test.

Exclusion Criteria. Not being able to drink, vomiting (more than twice within the prior 24 hours), recent history of seizures (1 or more in the previous 24 hours), alteration of the consciousness level, not being able to seat or stand up, signs of serious malaria (World Health Organization criteria), other chronic or severe diseases (i.e., cardiac, renal and hepatic diseases, HIV/AIDS, severe malnutrition), history of hypersensibility to any of the study drugs or drugs used as alternative treatment (i.e. mefloquine, artesunate, quinine or tetracycline/clindamycin), and suspicion of pregnancy or pregnancy (based on a urine pregnancy test).

Study arms and treatments. Two study arms were considered: Group 1 received the combination AQ+AS (COARSUCAM®) which was administered orally at an initial dose of 2 tablets (200 mg AQ/540 mg AS) followed by 2 additional doses of 2 tablets at 24 and 48 hours (6 tablets in 48 hours).

Group 2 received the combination Artemeter+lumefantrina (COARTEM®) administered orally at an initial dose of 4 tablets (80 mg artemeter/480 mg lumefantrina) followed by 5 additional doses of 4 tablets at 8, 24, 36, 48, and 60 hours (24 tablets in 60 hours)

Sample size. The sample size was estimated based on the expected proportion of failures for each one of the treatments in this population. Assuming a similar efficacy for both treatments (7) and considering a proportion of failures to treatment of 5% (range 1-11%) in a population of infinite size, a 5% significance level and a maximum tolerable error of +4%, a total of 100 study subjects are required to be included in each group. If 5% of the study subjects are lost in a 28 days study, a total of 105 will be needed in each group. All included subjects signed the Informed Consent.

Randomization. The assignment of treatments was made through a negative coordinated type sampling scheme (7) which consists in generating a list of randomized numbers from a normal distribution [0,1] and order the study subjects regarding this new list. These ordered study subjects were systematically chosen (in this case applying a ½ sampling fraction, i.e., 1 of every two for each treatment arm, since there were two arms) with an initial number randomly generated through a Bernoulli distribution. This process ensures a balanced allocation to the study arms.

Main outcomes. failure to take the drug on any of the first three days, parasitemia on day 2 greater than that on day 0, presence of parasitemia on day 7, diagnosis of severe malaria at any point after day 0, recurrent parasitemia after day 7 up to day 28 (8-11).

Analysis. Data were double-entered, and validated using Epi info© 2000 and the analysis was done using Stata™ 10.0. Per protocol analysis included patients who were properly randomised, had received the study drugs according to the protocol, and for whom data were available on the primary end point. All statistical tests were two-sided and an α-level <0.05 was considered a statistically significant result. For comparisons of continuous variables between groups, the t-test was used and for comparisons between more than two groups, one-way analysis of variance was used after assuring normality and homogeneity of variances assumptions were satisfied. For comparison of categorical variables, the chi-square test was used with the exact extension invoked when there were small numbers in the cells. The end points were any of the following: failure to take the drug on any of the first three days, parasitaemia on day 2 greater than that on day 0, presence of parasitaemia on day 7, diagnosis of severe malaria at any point after day 0, recurrent parasitaemia after day 7 up to day 28.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* fever (axillary temperature >37.5º C) or history of fever during the prior 48 hours in absence of another obvious cause (such as pneumonia, otitis media)
* a non-mixed P. falciparum infection with 250 and 100,000 asexual parasites/µl to be determined by a thick film or thick film and blood smear microscopic test

Exclusion Criteria:

* Not being able to drink
* vomiting (more than twice within the prior 24 hours)
* recent history of seizures (1 or more in the previous 24 hours)
* alteration of the consciousness level
* not being able to seat or stand up, signs of serious malaria (World Health Organization criteria)
* other chronic or severe diseases (i.e., cardiac, renal and hepatic diseases, HIV/AIDS, severe malnutrition)
* history of hypersensibility to any of the study drugs or drugs used as alternative treatment (i.e. mefloquine, artesunate, quinine or tetracycline/clindamycin)
* suspicion of pregnancy or pregnancy (based on a urine pregnancy test).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2008-09; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint was the adequate clinical and parasitological response (ACPR) | 28 days
  Absence of parasitemia on day 28, irrespective of axillary temperature, in patients who did not previously meet any of the criteria of early treatment failure, late clinical failure or late parasitological failure

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro AR Rico, Epidemiologist, Study Chair — Universidad Nacional de Colombia; Fernando FH De la Hoz, PhD, Principal Investigator — Universidad Nacional de Colombia; Alexandra AP Porras, Epidemiologist, Study Director — Universidad Nacional de Colombia; Freddy FC Cordoba, Epidemiologist, Study Chair — Chocó
Locations (1):
- San Rafael Hospital in Quibdó Chocó, Quibdó, Departamento del Chocó, Colombia